CLINICAL TRIAL: NCT03403842
Title: Treatment of Acute Post-operative Pain in Patients Undergoing Laparoscopic Colon Resections
Brief Title: Acute Post-operative Pain in Colon Resections
Acronym: ERAS-PO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Gemma, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 125/INT/2017
Record Dates: First submitted 2017-12-29; First posted 2018-01-19 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PERIDURAL (Active Comparator): Peridural catheter positioning with a continuous infusion of ropivacaine 0,2% 99 ml+ sufentanil 50 mcg at an infusion rate of 4-6 ml/h
  Interventions: Device: Peridural catheter
- PCA MORPHINE (Active Comparator): Patient controlled analgesia of endovenous morphine, injection dose 1 mg, lock-out time 10 minutes, maximum dosage for hour 4 mg
  Interventions: Drug: PCA Morphine
- SSTS (Experimental): Patients controlled analgesia of sublingual sufentanil tablet system, 15 mcg sufentanil tablets, lock out time 20 minutes
  Interventions: Device: Sublingual sufentanil tablet system

INTERVENTIONS:
Device: Sublingual sufentanil tablet system — Administration of sublingual sufentanil with a PCA
  Other Names: Zalviso
  Arms: SSTS
Device: Peridural catheter — Positioning of a peridural catheter with a continuous infusion of ropivacaine 0,2% 99 ml+sufentanil 50 mcg
  Arms: PERIDURAL
Drug: PCA Morphine — Administration of endovenous morphine with a PCA
  Arms: PCA MORPHINE

SUMMARY:
Objective of the study is to compare three different analgesic techniques in patients undergoing laparoscopic colon resections: peridural catheter, patient controlled analgesia of endovenous morphine and patient controlled analgesia of sufentanil sublingual tablets.

DETAILED DESCRIPTION:
159 patients undergoing laparoscopic colon resections will be enrolled and randomized in three different groups.

Patients in the first group will be subjected to the positioning of a peridural catheter with a continuous infusion of ropivacaine 0,2%99 ml+sufentanil 50 mcg at an infusion rate of 4-6 ml/h.

In the second group participants will receive an intraoperative bolus of morphine (0,05mg/kg) and post-operatively a patient controlled analgesia of endovenous morphine (injection dose 1 mg,lock-out 10 minutes,maximum morphine dosage for hour 4 mg).

In the third group the investigators will adopt an intraoperative bouls of morphine (0,05mg/kg) and post-operatively a patient controlled analgesia of sufentanil sublingual tablets( 15 mcg, lock-out 20 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Age>18 Patients undergoing laparoscopic colon resections/ Acceptance informed consent

Exclusion Criteria:

* Contraindications to the positioning of a peridural catheter/ Previous allergic reactions to the drugs used in the study/ inability of using patient controlled analgesia system

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity change in the post-operative period depending on the adopted analgesic treatment | NRS will be evaluated in recovery room at 30 minutes after the end of surgery and at 6-24-48-72 hours after the end of surgery or until to the end of the proposed analgesic treatment
  The intensity of acute post-operative pain will be evaluated ,according NRS(numerical rating scale) by our Acute pain Service.NRS is a 11 point scale for patient self-reporting of pain, where zero represents no pain and ten is considered as the worst pain ever possible

SECONDARY OUTCOMES:
Side effects | The onset of possible side effects will be monitored from randomization until to the end of the proposed analgesic treatment, assessed up to 72 hours
  Evaluation of possible side effects according to the technique adopted

CONTACTS AND LOCATIONS:
Locations (1):
- S. Raffaele Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feldheiser A, Aziz O, Baldini G, Cox BP, Fearon KC, Feldman LS, Gan TJ, Kennedy RH, Ljungqvist O, Lobo DN, Miller T, Radtke FF, Ruiz Garces T, Schricker T, Scott MJ, Thacker JK, Ytrebo LM, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 2: consensus statement for anaesthesia practice. Acta Anaesthesiol Scand. 2016 Mar;60(3):289-334. doi: 10.1111/aas.12651. Epub 2015 Oct 30. PMID 26514824
- [Background] Borzellino G, Francis NK, Chapuis O, Krastinova E, Dyevre V, Genna M. Role of Epidural Analgesia within an ERAS Program after Laparoscopic Colorectal Surgery: A Review and Meta-Analysis of Randomised Controlled Studies. Surg Res Pract. 2016;2016:7543684. doi: 10.1155/2016/7543684. Epub 2016 Aug 24. PMID 27642630
- [Background] Hubner M, Blanc C, Roulin D, Winiker M, Gander S, Demartines N. Randomized clinical trial on epidural versus patient-controlled analgesia for laparoscopic colorectal surgery within an enhanced recovery pathway. Ann Surg. 2015 Apr;261(4):648-53. doi: 10.1097/SLA.0000000000000838. PMID 25119117
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Frampton JE. Sublingual Sufentanil: A Review in Acute Postoperative Pain. Drugs. 2016 Apr;76(6):719-29. doi: 10.1007/s40265-016-0571-6. PMID 27067596